CLINICAL TRIAL: NCT07114354
Title: Enhancing Utility of Neuropsychological Evaluation for Earlier and Effective Diagnosis of Dementia in Parkinson's Disease
Acronym: PDCogniCare
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Queensland (Other)
Collaborators: Medical Research Future Fund (Other); Metro South Health (Other); Metro North Health (Unknown); Queensland University of Technology (Other); University of Sydney (Other); OPN365 (Unknown); Australian Dementia Network (Unknown); Dementia Australia (Unknown); Lions Club of Brisbane Inner North (Unknown); Parkinson's Queensland (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: HREC/2023/MNHA/100098
Record Dates: First submitted 2025-08-03; First posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-07

CONDITIONS: Dementia (Diagnosis); Parkinson Disease Dementia (PDD); Parkinson Disease (PD)
Keywords: Parkinson's disease; Dementia; Cognitive evaluation; Implementation
MeSH Terms: conditions — Dementia; Disease; Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PDCogniCare (Other): All eligible people living with Parkinson's disease who consent to participate will be registered into the PDCogniCare platform.
  Interventions: Other: PDCogniCare platform

INTERVENTIONS:
Other: PDCogniCare platform — Digital platform designed to support early and accurate detection of dementia in people living with Parkinson's disease

SUMMARY:
Dementia is observed in 80% of people living with advanced stage Parkinson's disease, however, there are inadequate opportunities for early and effective diagnosis of dementia in current clinical practice. This study aims to identify whether a new tool called PDCogniCare, can improve detection of dementia in people living with Parkinson's disease, and to explore what factors might influence its use in healthcare services.

DETAILED DESCRIPTION:
The PDCogniCare tool integrates best practice guidelines for cognitive evaluations in people living with Parkinson's disease, along with a tailored digital platform to support guideline implementation and routinely track cognitive changes throughout the disease course. We hypothesize that PDCogniCare will significantly enhance cognitive evaluations within healthcare services. Embedded process and economics evaluations will inform implementation and sustainable business models of PDCogniCare.

ELIGIBILITY:
Inclusion Criteria:

* People living with idiopathic Parkinson's disease, one year or more post-diagnosis, attending Movement Disorder Clinics

Exclusion Criteria:

* People with severe Parkinson's disease who aren't able to communicate
* People with comorbid neurological conditions (e.g. Stroke)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 275 (Estimated)
Dates: Start 2025-08-18 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in percentage of people with Parkinson's disease diagnosed with dementia | 12 months from enrolment

SECONDARY OUTCOMES:
Change in percentage of people with Parkinson's disease diagnosed with mild cognitive impairment | 12 months from enrolment

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pourzinal D, King J, Sivakumaran K, Yang J, McCann E, Mitchell LK, Brooks D, Lehn A, Liddle J, Pachana NA, Tinson H, Shrubsole K, Bailey DX, Dissanayaka NN. Evaluating evidence for a neuropsychological toolkit to predict cognitive decline in PD: A systematic review. Clin Neuropsychol. 2025 Jun 4:1-28. doi: 10.1080/13854046.2025.2511966. Online ahead of print. PMID 40464273
- [Background] Pourzinal D, Elgey C, Bailey DX, Yang J, Lehn A, Tinson H, Liddle J, Brooks D, Naismith SL, Shrubsole K, Marsh R, Mitchell LK, Pachana NA, King J, Dissanayaka NN. Diagnosis, evaluation & management of cognitive disorders in Parkinson's disease: A systematic review. Int Psychogeriatr. 2025 May 12:100081. doi: 10.1016/j.inpsyc.2025.100081. Online ahead of print. PMID 40360335